CLINICAL TRIAL: NCT07148648
Title: Institutional Experience With Chest Wall Reconstruction Using Sternal Steel Wires: A Case Series Study
Status: Completed | Type: Observational
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principal Investigator, University of Health Sciences Lahore
Other Study IDs: IRB/2025/1653/SIMS
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chest Wall Mechanics; Chest Wall Deformity; Chest Wall Tumor; Chest Wall Disease
Keywords: sternal steel wires; chest wall reconstruction; respiratory mechanics; flail segment; chest wall tumors; chest wall resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wires Group: all the participants who undergo chest wall reconstruction using sternal steel wires, number 05 are included in this group.
  Interventions: Procedure: Chest Wall Reconstruction

INTERVENTIONS:
Procedure: Chest Wall Reconstruction — there are many methods described in literature for reconstruction of chest wall after chest wall resection. The investigators are focusing on chest wall reconstruction using steel wires in this study.

SUMMARY:
Chest wall resections, often performed for tumors, infections, or trauma, result in significant defects that require reconstruction to restore structural integrity and functionality. The use of twisted stainless steel wires (No. 05) for chest wall reconstruction offers a cost-effective and practical alternative. Steel wires provide robust structural support, allow dynamic movement of the chest wall during respiration, and are associated with improved postoperative pain control.

DETAILED DESCRIPTION:
The chest wall, a complex dynamic structure composed of both rigid and soft tissues, plays a vital role in protecting thoracic organs and maintaining the mechanics of respiration. Reconstruction following chest wall resection is critical not only to achieve defect closure but also to preserve respiratory mechanics and minimize postoperative complications. The primary goals include providing structural support, ensuring stability, and achieving soft tissue coverage while maintaining chest wall flexibility and minimizing pain. Chest wall reconstruction using sternal steel wires enable better chest wall recoil, which is crucial for maintaining normal respiratory mechanics. Additionally, studies suggest that the use of steel wires reduces the incidence of chronic pain, as they do not involve direct exposure to synthetic materials that could irritate surrounding tissues or provoke inflammatory responses. The affordability and simplicity of steel wire-based reconstruction make it particularly suitable for underserved populations in Pakistan, where healthcare resources are limited, and the majority of patients cannot afford expensive surgical materials.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing chest wall resection due to tumors or trauma.

Exclusion Criteria:

* Patients with contraindications to General Anesthesia.
* Patients having chest wall infection.
* Patients with pre-existing chest wall deformities or severe chronic respiratory diseases.
* Patients who undergo reoperation or develop intraoperative complications affecting the chest wall reconstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants diagnosed with conditions requiring chest wall reconstruction and admitted to the thoracic surgery ward, emergency department, or outpatient department during the study period will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Chest Wall Recoil | 30 days post-operatively
  Chest wall recoil after reconstruction is defined as maintenance of normal chest wall movement during respiration without paradoxical motion.
  It is assessed using spirometry (Forced Vital Capacity [FVC] and Forced Expiratory Volume in 1 second [FEV1]) compared with baseline/preoperative predicted values, radiological evaluation (postoperative chest X-rays for symmetrical expansion) and clinical observation (absence of paradoxical chest wall movement on examination).
  Preserving chest wall recoil is essential for normal breathing mechanics. Reconstruction with sternal steel wires aims to restore physiological elasticity, maintain ventilatory efficiency, and reduce respiratory complications.

SECONDARY OUTCOMES:
Post-Operative Pain Control | 24 hours, 72 hours and 07 days
  Post-operative pain control is measured using the Visual Analogue Scale (VAS) ranging from 0 (no pain) to 10 (worst imaginable pain). It is recorded at 24 hours, 72 hours, and 7 days postoperatively.
  Pain is a critical determinant of recovery, respiratory function, and overall patient satisfaction. Evaluating pain scores will help determine whether sternal steel wire fixation provides a less painful and more tolerable method of chest wall reconstruction compared to alternative techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Professor Of Thoracic Surgery, Principal Investigator — Services Institute Of Medical Sciences (SIMS), Services Hospital, Lahore
Locations (1):
- Services Institute Of Medical Sciences (SIMS), Services Hospital, Lahore, Lahore, Punjab Province, Pakistan